CLINICAL TRIAL: NCT00960739
Title: Phase II Study of the Association of Iodobenzylguanidine Meta-I131 (I131 MIBG) and Topotecan in the Treatment of Refractory or Relapsed Metastatic Neuroblastoma
Brief Title: Iodobenzylguanidine Meta-I131 and Topotecan in Young Patients With Refractory or Relapsed Metastatic Neuroblastoma
Acronym: MIITOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIITOP-0607
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized unresectable neuroblastoma; recurrent neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Topotecan; Hematopoietic Stem Cell Transplantation; 3-Iodobenzylguanidine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topotecan / 131-iodine MIBG association (Experimental): * The topotecan hydrochloride is administered intravenously over five days to dose of 0.7 mg/ m²/day from day 1 to day 5 (first cycle), then from day 21 to day 25 (second cycle). *
  * Iobenguane I 131: 444 MBq / kg of 131-iodine MIBG is administered on day 1 with activity up to 11,100 MBq per injection. *
  * A dosimetry is performed during hospitalization.
  * A second dose of 131-iodine MIBG (maximum 11 100 MBq) is administered to D21 so as to obtain a total body irradiation of 4 Gy. *
  * Autologous hematopoietic stem cell transplantation : Hematopoietic stem cells are reinjected 10 days after the second injection of 131-iodine MIBG.
    * If the dose of total-body irradiation of 4 Gy is reached during the first cycle, the second cycle is canceled.
  Interventions: Drug: Topotecan hydrochloride; Procedure: Autologous hematopoietic stem cell transplantation; Radiation: iobenguane I 131; Radiation: total-body irradiation

INTERVENTIONS:
Drug: Topotecan hydrochloride — The topotecan hydrochloride is administered intravenously over five days to dose of 0.7 mg/ m²/day from day 1 to day 5 (first cycle), then from day 21 to day 25 (second cycle)
  Other Names: Topotecan
Procedure: Autologous hematopoietic stem cell transplantation — Hematopoietic stem cells are reinjected 10 days after the second injection of 131-iodine MIBG
  Other Names: hematopoietic stem cell transplantation
Radiation: iobenguane I 131 — 444 MBq / kg of 131-iodine MIBG is administered on day 1 with activity
Radiation: total-body irradiation — the dose of total-body irradiation of 4 Gy is reached during the first cycle, the second cycle is canceled (131-iodine MIBG and Topotecan)

SUMMARY:
RATIONALE: Radioactive drugs, such as iodobenzylguanidine meta-I131, may carry radiation directly to tumor cells and not harm normal cells. Drugs used in chemotherapy, such as topotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. A stem cell transplant may be able to replace the cells that were destroyed by iodobenzylguanidine meta-i131 and topotecan hydrochloride.

PURPOSE: This phase II trial is studying the side effects of iodobenzylguanidine meta-I131 given together with topotecan hydrochloride and to see how well it works in treating young patients with refractory or relapsed metastatic neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of iodobenzylguanidine meta-I131 (^131I-MIBG) and topotecan in young patients with refractory or relapsed metastatic neuroblastoma.

Secondary

* Determine the hematological and extra-hematological toxicities of this regimen.

OUTLINE: This is a multicenter study.

During the 21 days before treatment begins, autologous peripheral blood stem cells (PBSC) are collected.

Patients receive topotecan hydrochloride IV over 30 minutes daily on days 1-5 and iodobenzylguanidine meta-^131I IV over 2 hours on day 1. Treatment repeats every 21 days for 2 courses. Patients also undergo total-body irradiation.

On day 10 of the second course, autologous PBSC are reinfused.

After completion of study therapy, patients are followed at 6 and 12 months.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed neuroblastoma
* Metastatic disease that is recurrent or refractory to induction therapy
* Primary or metastatic tumor target with MIBG fixation (tumor/soft tissue) > 2
* Autologous bone marrow or peripheral blood stem cells must be available
* WHO performance status (PS) 0-1 OR Lansky PS 70-100%
* Life expectancy > 2 months
* ANC ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine clearance normal for age
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior hypersensitivity to topotecan or its excipients
* No toxicity to other organs ≥ NCI-CTCAE v3.0 grade 2
* No other debilitating disease
* No HIV positivity
* More than 30 days since prior external-beam radiation (6 weeks if cranio-spinal, abdominal, or pulmonary)
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas)
* No other contraindicated biologic therapy that cannot be discontinued for ≥ 4 courses during MIBG therapy

Exclusion criteria:

* Pregnancy or breastfeeding women
* HIV positive
* Participation to another phase I,II or III clinical trial
* Other invalidating pathology
* Concomitant treatment interfering with MIBG
* Hypersensibility to Topotecan

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 12 months

SECONDARY OUTCOMES:
Toxicity | Up to 30 days after study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie Defachelles, MD, Principal Investigator — Centre Oscar Lambret
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital des Enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sevrin F, Kolesnikov-Gauthier H, Cougnenc O, Bogart E, Schleiermacher G, Courbon F, Gambart M, Giraudet AL, Corradini N, Badel JN, Rault E, Oudoux A, Deley MCL, Valteau-Couanet D, Defachelles AS. Phase II study of 131 I-metaiodobenzylguanidine with 5 days of topotecan for refractory or relapsed neuroblastoma: Results of the French study MIITOP. Pediatr Blood Cancer. 2023 Nov;70(11):e30615. doi: 10.1002/pbc.30615. Epub 2023 Aug 13. PMID 37574821